CLINICAL TRIAL: NCT03343457
Title: A Randomized Intervention and Coordination Program Aiming at Return To Work for Women With Long Term Sick Leave
Brief Title: Return To Work for People on Long Term Sick Leave
Acronym: Vitalis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VITALIS 2010
Record Dates: First submitted 2017-10-30; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Anxiety; Chronic Pain
Keywords: Anxiety; Chronic Pain
MeSH Terms: conditions — Anxiety Disorders; Chronic Pain | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acceptance Commitment Therapy (Experimental): Acceptance Commitment Therapy. Cognitive therapy
  Interventions: Behavioral: Cognitive therapy
- Multidisciplinary assessment (Experimental): Assessment of a team. Cognitive therapy
  Interventions: Behavioral: Cognitive therapy
- Control (No Intervention): Control group

INTERVENTIONS:
Behavioral: Cognitive therapy
  Other Names: ACT, multidisciplinary assessment
  Arms: Acceptance Commitment Therapy; Multidisciplinary assessment

SUMMARY:
Vitalis was a randomized controlled intervention study that addressed women on long-term sick leave in Uppsala County. Participants were on sick leave due to mental illness and/or pain and were expected to reach the time limit within the in health insurance. Of the total of 947 eligible reaching the time limit during 2010-2012 648 persons met the projects inclusion- and exclusion criteria and were invited to participate. Of these, 327 persons (50.4%) gave informed consent and was thereafter randomly assigned one of the following groups: 1) multimodal treatment team (TEAM) 2) psychotherapy with Acceptance and Commitment Therapy (ACT), or 3) control group. The main purpose of the study was to facilitate the return to work (preventing a return to the public health insurance) and to improve participants' health during the project period of one year.

DETAILED DESCRIPTION:
Vitalis was a randomized controlled intervention study that addressed women on long-term sick leave in Uppsala County. Participants were on sick leave due to mental illness and/or pain and were expected to reach the time limit within the in health insurance. Of the total of 947 eligible reaching the time limit during 2010-2012 648 persons met the projects inclusion- and exclusion criteria and were invited to participate. Of these, 327 persons (50.4%) gave informed consent and was thereafter randomly assigned one of the following groups: 1) multimodal treatment team (TEAM) 2) psychotherapy with Acceptance and Commitment Therapy (ACT), or 3) control group. The main purpose of the study was to facilitate the return to work (preventing a return to the public health insurance) and to improve participants' health during the project period of one year.

The participants of the TEAM group received individual meetings/assessments with a doctor, psychologist, occupational therapist and social worker, each assessing the participant's problems in relation to the return to work goal. The TEAM then worked out an individualized plan of actions/treatments, which then was presented to the participant. Suggested and accepted actions were psychotherapy (60%, average 9.2 sessions); Occupational Therapist (72%, average 3.7 sessions); social worker (36%, average 6.5 sessions) and further medical investigations/referrals initiated by physicians (41%).

In the ACT group all participants received psychotherapy with ACT with an average of 10.0 sessions (range 1-23) during the project year.

In addition to the medical assessment/treatments all participants in the intervention groups also participated in scheduled collaboration meetings with representatives from the health insurance agency and employment office in order to establish an agreement and justification on the rehabilitation goals. The participant and a health professional from the project participated in these collaborations meetings.

During the project year the participants filled in questionnaire at three points in time in which they rated their views on returning to work as well as various aspects of their health. Data whether the participants had returned to the health insurance as well as the number of reimbursed days during the first years, was collected from the health insurance register after one year.

ELIGIBILITY:
Inclusion Criteria:

* On sick leave for mental illness and/or chronic pain

Exclusion Criteria:

* High risk for suicide
* Ongoing alcohol/substance abuse
* Major mental illness (schizophrenia, bipolar disorder type I, severe social dysfunction/personality disorder)
* Participation in psychotherapy or another vocational rehabilitation program.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2012-12-31 (Actual)

PRIMARY OUTCOMES:
Return to work (RTW) | One year
  Return to work measured as self-reported change in working hours

REFERENCES:
- [Derived] Berglund E, Anderzen I, Helgesson M, Lytsy P, Andersen A. Work participation after receiving multidisciplinary treatment or acceptance and commitment therapy intervention for return to work: long-term follow-up of a randomized controlled trial among sick-listed individuals with mental disorders and/or chronic pain. BMC Public Health. 2024 Dec 21;24(1):3558. doi: 10.1186/s12889-024-21116-1. PMID 39709368